CLINICAL TRIAL: NCT00362115
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Dose-Ranging Study of the Efficacy, Safety and Tolerability of TAK-491 in Subjects With Mild to Moderate Uncomplicated Essential Hypertension
Brief Title: Safety and Efficacy of Azilsartan Medoxomil in Participants With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-491-005; U1111-1113-8783 (Registry Identifier: WHO)
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure; diastolic blood pressure; drug therapy
MeSH Terms: conditions — Hypertension | interventions — azilsartan medoxomil; azilsartan; olmesartan; Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Azilsartan Medoxomil 5 mg QD (Experimental)
  Interventions: Drug: Azilsartan Medoxomil
- Azilsartan Medoxomil 10 mg QD (Experimental)
  Interventions: Drug: Azilsartan Medoxomil
- Azilsartan Medoxomil 20 mg QD (Experimental)
  Interventions: Drug: Azilsartan Medoxomil
- Azilsartan Medoxomil 40 mg QD (Experimental)
  Interventions: Drug: Azilsartan Medoxomil
- Azilsartan Medoxomil 80 mg QD (Experimental)
  Interventions: Drug: Azilsartan Medoxomil
- Olmesartan 20 mg QD (Active Comparator)
  Interventions: Drug: Olmesartan
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azilsartan Medoxomil — Azilsartan medoxomil 5 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 5 mg QD
Drug: Azilsartan Medoxomil — Azilsartan medoxomil 10 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 10 mg QD
Drug: Azilsartan Medoxomil — Azilsartan medoxomil 20 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 20 mg QD
Drug: Azilsartan Medoxomil — Azilsartan medoxomil 40 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 40 mg QD
Drug: Azilsartan Medoxomil — Azilsartan medoxomil 80 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 80 mg QD
Drug: Olmesartan — Olmesartan 20 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
  Other Names: Benicar
  Arms: Olmesartan 20 mg QD
Drug: Placebo — Matching placebo tablets, orally, once daily for up to 8 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and tolerability of azilsartan medoxomil, once daily (QD), in individuals with hypertension.

DETAILED DESCRIPTION:
Hypertension affects approximately 50 million individuals in the United States. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. Data from the Framingham Heart study suggest that the lifetime risk of developing hypertension among 55- to 65-year-old individuals is greater than 90%. According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. Despite the availability of hypertension treatments, hypertension remains inadequately controlled; only about one third of patients continue to maintain control successfully. To help address these matters, the Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure proposes a more aggressive intervention to hypertension management with more potent antihypertensive agents and combination therapy.

Takeda Global Research & Development Center, Inc. is developing TAK-491 (azilsartan medoxomil) to treat mild to moderate essential hypertension. Azilsartan medoxomil is a prodrug that is rapidly hydrolyzed to the activity moiety, azilsartan, which is an angiotensin II type 1 receptor antagonist. This study is proposed to evaluate the efficacy, safety and tolerability of multiple doses of azilsartan medoxomil at five dose levels in subjects with mild to moderate uncomplicated essential hypertension.

Individuals who want to participate in this study will be required to provide written informed consent. Study participation is anticipated to be about 11 weeks. Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, vital signs including sitting and standing blood pressure and pulse, body height and weight, physical examinations, electrocardiogram Outside of the study center, participants will be required to wear an ambulatory blood pressure monitoring device at approximately 24 and 36 hour intervals.

ELIGIBILITY:
Inclusion Criteria

1. Mild to moderate uncomplicated essential hypertension.
2. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
3. Must be in good health as determined by a physician.
4. The subject has clinical laboratory evaluations within the reference range for the testing laboratory unless the results are deemed not clinically significant by the investigator or sponsor.
5. The subject is willing to discontinue current antihypertensive medications at Screening Day minus 21.

Exclusion Criteria

1. Diastolic blood pressure less than 95 or greater than 114 mmHg at Placebo Run-in Day minus 14 or Randomization visit, or systolic blood pressure greater than 180 mm Hg.
2. Decrease of more than or equal to 8 mm Hg in clinic diastolic blood pressure between Placebo Run-in Day minus 14 and Randomization visit.
3. Has taken within 7 days prior to placebo run-in, or is expected to take medications known to affect blood pressure and is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:
4. Hypersensitive to angiotensin II receptor blockers.
5. History of an acute myocardial infarction within 12 months prior to Screening, history of coronary revascularization within 6 months prior to Screening, or any history of heart failure, post-myocardial infarction angina, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
6. Clinically significant cardiac conduction defects (eg, 3rd degree atrioventricular block, left bundle branch block, atrial fibrillation or flutter).
7. Secondary hypertension of any etiology.
8. Upper arm circumference less than 24 or greater than 42 cm.
9. Works night (3rd) shift (defined as 11pm to 7am).
10. Non-compliant (less than 80%) with study medication during Placebo Run-in period.
11. Significant, moderate to severe renal dysfunction (confirmed by serum creatinine of greater than 2 mg per dl or disease (including renal artery stenosis or known nephrotic proteinuria).
12. History of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within the past 2 years.
13. Previous history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not include those subjects with basal cell or Stage 1 squamous cell carcinoma of the skin).
14. Type 1 or uncontrolled type 2 diabetes mellitus (confirmed by glycosylated hemoglobin greater than 9.5%).
15. Alanine transaminase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
16. Currently is participating in another investigational study or has participated in an investigational study within 30 days prior to randomization.
17. Any other serious disease or condition at Screening (or randomization) that would compromise subject safety, might affect life expectancy, or make it difficult to successfully manage and follow the subject according to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2006-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (54):
- United States (46):
  - Huntsville, Alabama
  - Ozark, Alabama
  - Mesa, Arizona
  - Little Rock, Arkansas
  - Carmichael, California
  - Long Beach, California
  - San Diego, California
  - Tustin, California
  - Denver, Colorado
  - Stamford, Connecticut
  - Trumbull, Connecticut
  - Waterbury, Connecticut
  - Hollywood, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Atlanta, Georgia
  - Evansville, Indiana
  - Shawnee Mission, Kansas
  - Auburn, Maine
  - Trenton, New Jersey
  - Binghamtom, New York
  - Rochester, New York
  - Burlington, North Carolina
  - Charlotte, North Carolina
  - Concord, North Carolina
  - Hickory, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Anderson, South Carolina
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Euless, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Lakewood, Washington
  - Renton, Washington
  - Madison, Wisconsin
- Argentina (3):
  - BA
  - Córdoba
  - Ushuaia
- Mexico (4):
  - Guadalajara, Jal
  - Mexico City
  - Monterrey Nuevo Leon
  - Morelia, Michoacan
- Lima, Peru

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 76 investigative sites in Argentina, Mexico, Peru and the United States from 16 May 2006 to 07 December 2006.
Pre-assignment Details: Participants with mild to moderate uncomplicated essential hypertension were enrolled in one of seven, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 5 mg QD: Azilsartan medoxomil 5 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 10 mg QD: Azilsartan medoxomil 10 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 20 mg QD: Azilsartan medoxomil 20 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 40 mg QD: Azilsartan medoxomil 40 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
- Azilsartan Medoxomil 80 mg QD: Azilsartan medoxomil 80 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
- Olmesartan 20 mg QD: Olmesartan 20 mg and comparator matching placebo tablets, orally, once daily for up to 8 weeks.
- Placebo QD: Matching placebo tablets, orally, once daily for up to 8 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Started | 65 | 65 (1 participant failed to receive double-blind medication.) | 64 | 63 (1 participant failed to receive double-blind medication.) | 64 | 64 (1 participant failed to receive double-blind medication.) | 64 (1 participant failed to receive double-blind medication.)
Completed | 63 | 59 | 57 | 59 | 57 | 57 | 52
Not Completed | 2 | 6 | 7 | 4 | 7 | 7 | 12
Not completed — Adverse Event | 0 | 1 | 1 | 1 | 2 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 1 | 0 | 1 | 3 | 4
Not completed — Lack of Efficacy | 1 | 0 | 5 | 2 | 2 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Other | 0 | 1 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD | Total
Number analyzed (Participants) | 65 | 63 | 64 | 62 | 64 | 63 | 61 | 442
Age Categorical [Number; unit: participants]
  <45 years | 12 | 5 | 10 | 9 | 12 | 10 | 11 | 69
  Between 45 and 64 years | 45 | 52 | 46 | 43 | 41 | 46 | 36 | 309
  ≥65 years | 8 | 6 | 8 | 10 | 11 | 7 | 14 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 30 | 33 | 28 | 34 | 32 | 218
  Male | 36 | 31 | 34 | 29 | 36 | 29 | 29 | 224

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sitting Clinic Diastolic Blood Pressure.
Description: The change in sitting clinic diastolic blood pressure measured at final visit or week 8 relative to baseline. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 8.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 63 | 63 | 63 | 61 | 63 | 63 | 58
mmHg | -10.8 (1.08) | -13.1 (1.08) | -11.5 (1.08) | -13.6 (1.10) | -11.6 (1.08) | -11.0 (1.08) | -7.9 (1.12)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0631, ANCOVA — P-value from analysis of covariance with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value is presented; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-5.96 to 0.16]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0008, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-8.33 to -2.20]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0188, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-6.73 to -0.61]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-8.80 to -2.63]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0177, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-6.77 to -0.65]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.8550, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI [-2.72 to 3.27]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1719, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-5.08 to 0.91]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.7469, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-3.49 to 2.50]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-5.55 to 0.49]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.7294, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-3.52 to 2.47]

2. Secondary Outcome: Change From Baseline in Sitting Clinic Systolic Blood Pressure.
Description: The change in sitting clinic systolic blood pressure measured at final visit or week 8 relative to baseline. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 8
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 63 | 63 | 63 | 61 | 63 | 63 | 58
mmHg | -11.0 (1.66) | -15.7 (1.66) | -14.7 (1.66) | -17.1 (1.69) | -13.3 (1.66) | -13.5 (1.66) | -4.9 (1.73)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0111, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-10.84 to -1.41]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.8, 95% CI 2-sided [-15.51 to -6.08]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.8, 95% CI 2-sided [-14.53 to -5.10]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.3, 95% CI 2-sided [-17.02 to -7.52]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0005, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-13.19 to -3.76]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2768, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-2.06 to 7.17]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3688, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-6.74 to 2.51]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.6293, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -1.1, 95% CI 2-sided [-5.75 to 3.48]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1298, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-8.25 to 1.06]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.9315, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-4.41 to 4.82]

3. Secondary Outcome: Change From Baseline in Standing Clinic Systolic Blood Pressure.
Description: The change in standing clinic systolic blood pressure measured at final visit or week 8 relative to baseline. Systolic blood pressure is the arithmetic mean of the 3 trough standing systolic blood pressure measurements.
Time Frame: Baseline and Week 8.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 63 | 63 | 63 | 61 | 62 | 63 | 58
mmHg | -11.4 (1.78) | -13.4 (1.78) | -16.1 (1.78) | -14.6 (1.81) | -14.0 (1.79) | -11.4 (1.78) | -3.3 (1.85)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0016, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.1, 95% CI 2-sided [-13.17 to -3.09]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.1, 95% CI 2-sided [-15.17 to -5.09]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.8, 95% CI 2-sided [-17.80 to -7.72]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-16.36 to -6.20]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.7, 95% CI 2-sided [-15.75 to -5.63]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.9909, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-4.96 to 4.91]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.4213, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-6.96 to 2.92]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0646, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.7, 95% CI 2-sided [-9.59 to 0.28]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2107, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-8.15 to 1.80]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3059, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-7.54 to 2.37]

4. Secondary Outcome: Change From Baseline in Standing Clinic Diastolic Blood Pressure.
Description: The change in standing clinic diastolic blood pressure measured at final visit or week 8 relative to baseline. Diastolic blood pressure is the arithmetic mean of the 3 trough standing diastolic blood pressure measurements.
Time Frame: Baseline and Week 8.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 63 | 63 | 63 | 61 | 62 | 63 | 58
mmHg | -9.2 (1.17) | -11.0 (1.18) | -10.2 (1.17) | -11.3 (1.19) | -11.2 (1.18) | -10.8 (1.17) | -6.9 (1.23)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.1653, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-5.69 to 0.98]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0151, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-7.50 to -0.81]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0480, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-6.70 to -0.03]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0098, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-7.81 to -1.08]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0113, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-7.68 to -0.98]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3416, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-1.68 to 4.84]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.8973, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-3.49 to 3.06]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.7292, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-2.69 to 3.84]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.7646, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-3.79 to 2.79]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.8133, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-3.67 to 2.88]

5. Secondary Outcome: Change From Baseline in 24-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean systolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 56 | 45 | 47 | 41 | 45 | 50 | 43
mmHg | -7.5 (1.34) | -12.1 (1.49) | -11.1 (1.46) | -15.8 (1.57) | -12.4 (1.49) | -9.3 (1.42) | 1.0 (1.53)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-12.51 to -4.51]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.1, 95% CI 2-sided [-17.31 to -8.90]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.1, 95% CI 2-sided [-16.27 to -7.95]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -16.8, 95% CI 2-sided [-21.07 to -12.46]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.4, 95% CI 2-sided [-17.58 to -9.17]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3735, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-2.10 to 5.58]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1668, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-6.91 to 1.20]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3629, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-5.86 to 2.15]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0022, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.5, 95% CI 2-sided [-10.67 to -2.36]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1303, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-7.18 to 0.93]

6. Secondary Outcome: Change From Baseline in 24-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 56 | 45 | 47 | 41 | 45 | 50 | 43
mmHg | -4.2 (0.90) | -7.3 (1.01) | -7.5 (0.99) | -9.6 (1.06) | -8.2 (1.01) | -6.2 (0.96) | 1.2 (1.03)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-8.12 to -2.72]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-11.33 to -5.65]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.7, 95% CI 2-sided [-11.52 to -5.90]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.8, 95% CI 2-sided [-13.73 to -7.91]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.5, 95% CI 2-sided [-12.31 to -6.64]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1249, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-0.56 to 4.61]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.4542, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-3.79 to 1.70]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3574, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.97 to 1.44]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0184, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-6.18 to -0.57]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1450, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-4.77 to 0.70]

7. Secondary Outcome: Change From Baseline in the 12-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean systolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 56 | 45 | 47 | 41 | 45 | 50 | 43
mmHg | -7.2 (1.54) | -13.0 (1.72) | -11.8 (1.68) | -17.2 (1.80) | -13.0 (1.72) | -7.4 (1.63) | 0.6 (1.76)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0009, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-12.46 to -3.26]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.6, 95% CI 2-sided [-18.46 to -8.77]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.4, 95% CI 2-sided [-17.21 to -7.63]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -17.9, 95% CI 2-sided [-22.83 to -12.92]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.7, 95% CI 2-sided [-18.52 to -8.84]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.9424, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-4.25 to 4.58]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0189, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-10.26 to -0.93]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0612, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-9.01 to 0.21]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.9, 95% CI 2-sided [-14.63 to -5.07]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0175, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-10.33 to -1.00]

8. Secondary Outcome: Change From Baseline in the 12-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 56 | 45 | 47 | 41 | 45 | 50 | 43
mmHg | -3.6 (1.05) | -7.3 (1.18) | -8.0 (1.15) | -10.0 (1.23) | -8.7 (1.18) | -5.1 (1.12) | 0.6 (1.21)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0108, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-7.26 to -0.95]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-11.16 to -4.55]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-11.82 to -5.26]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.6, 95% CI 2-sided [-13.98 to -7.20]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.2, 95% CI 2-sided [-12.52 to -5.90]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3060, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-1.45 to 4.59]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1823, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-5.37 to 1.02]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0751, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-6.01 to 0.29]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0034, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-8.18 to -1.64]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0306, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-6.72 to -0.33]

9. Secondary Outcome: Change From Baseline in the 10-12-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 10 to 12-hour mean systolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 10-12-hour mean is the average of all measurements recorded after dosing during these 2 hours.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 54 | 44 | 45 | 40 | 45 | 49 | 41
mmHg | -8.0 (1.93) | -11.4 (2.14) | -12.2 (2.12) | -17.4 (2.24) | -13.7 (2.12) | -7.8 (2.03) | 0.1 (2.22)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0061, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.1, 95% CI 2-sided [-13.90 to -2.33]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.5, 95% CI 2-sided [-17.56 to -5.44]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.3, 95% CI 2-sided [-18.34 to -6.28]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -17.5, 95% CI 2-sided [-23.75 to -11.34]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.8, 95% CI 2-sided [-19.86 to -7.80]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.9355, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-5.74 to 5.28]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2223, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-9.41 to 2.20]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1328, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-10.19 to 1.35]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0016, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.7, 95% CI 2-sided [-15.61 to -3.70]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0437, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-11.70 to -0.17]

10. Secondary Outcome: Change From Baseline in the 10-12-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 10 to 12-hour mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 10-12-hour mean is the average of all measurements recorded after dosing during these 2 hours.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 54 | 44 | 45 | 40 | 45 | 49 | 41
mmHg | -3.8 (1.37) | -5.7 (1.52) | -7.4 (1.50) | -9.1 (1.59) | -8.8 (1.50) | -4.7 (1.44) | 0.5 (1.58)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0417, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-8.39 to -0.16]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0053, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-10.44 to -1.84]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0004, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.8, 95% CI 2-sided [-12.12 to -3.56]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.6, 95% CI 2-sided [-13.97 to -5.16]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.3, 95% CI 2-sided [-13.60 to -5.03]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.6372, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-2.97 to 4.85]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.6588, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-5.05 to 3.20]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2082, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-6.72 to 1.47]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0437, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-8.57 to -0.12]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0495, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-8.19 to -0.01]

11. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean systolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 8
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 53 | 43 | 45 | 38 | 44 | 48 | 39
mmHg | -10.9 (1.78) | -14.9 (1.98) | -12.0 (1.93) | -18.8 (2.10) | -13.9 (1.95) | -13.8 (1.87) | -1.5 (2.08)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0007, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.4, 95% CI 2-sided [-14.74 to -3.97]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.4, 95% CI 2-sided [-19.02 to -7.73]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.4, 95% CI 2-sided [-16.00 to -4.83]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -17.3, 95% CI 2-sided [-23.11 to -11.47]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.4, 95% CI 2-sided [-18.01 to -6.78]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2594, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [-2.17 to 8.01]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.6859, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-6.46 to 4.26]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.4898, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-3.43 to 7.15]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0760, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-10.55 to 0.53]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.9647, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-5.44 to 5.21]

12. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 53 | 43 | 45 | 38 | 44 | 48 | 39
mmHg | -7.6 (1.27) | -11.3 (1.41) | -8.9 (1.38) | -14.0 (1.50) | -9.0 (1.39) | -9.6 (1.33) | -0.3 (1.48)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-11.13 to -3.43]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.0, 95% CI 2-sided [-15.01 to -6.97]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.6, 95% CI 2-sided [-12.59 to -4.64]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.6, 95% CI 2-sided [-17.79 to -9.50]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.7, 95% CI 2-sided [-12.69 to -4.70]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2790, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-1.63 to 5.62]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3772, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-5.53 to 2.10]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.7302, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-3.11 to 4.43]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0302, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-8.31 to -0.42]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.7644, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-3.22 to 4.38]

13. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 56 | 45 | 47 | 41 | 45 | 50 | 43
mmHg | -7.8 (1.43) | -13.0 (1.59) | -11.6 (1.56) | -17.3 (1.67) | -13.1 (1.59) | -8.6 (1.51) | 0.7 (1.63)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.4, 95% CI 2-sided [-12.70 to -4.19]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.7, 95% CI 2-sided [-18.19 to -9.24]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.2, 95% CI 2-sided [-16.66 to -7.80]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -17.9, 95% CI 2-sided [-22.51 to -13.35]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.7, 95% CI 2-sided [-18.21 to -9.25]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.6905, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-3.26 to 4.91]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0433, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-8.76 to -0.13]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1736, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-7.22 to 1.31]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.7, 95% CI 2-sided [-13.08 to -4.23]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0429, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-8.77 to -0.14]

14. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 56 | 45 | 47 | 41 | 45 | 50 | 43
mmHg | -4.2 (0.96) | -7.7 (1.07) | -8.0 (1.05) | -10.6 (1.12) | -8.7 (1.07) | -6.0 (1.01) | 0.7 (1.09)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0009, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-7.77 to -2.04]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.3, 95% CI 2-sided [-11.33 to -5.32]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.7, 95% CI 2-sided [-11.63 to -5.67]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-14.34 to -8.18]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.4, 95% CI 2-sided [-12.37 to -6.36]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2068, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-0.98 to 4.50]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2622, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-4.56 to 1.25]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1730, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-4.85 to 0.88]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0025, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-7.56 to -1.62]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0681, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-5.60 to 0.20]

15. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 54 | 44 | 46 | 39 | 44 | 49 | 40
mmHg | -7.3 (1.56) | -11.1 (1.73) | -10.4 (1.69) | -13.1 (1.83) | -11.4 (1.72) | -10.6 (1.63) | 1.3 (1.81)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0004, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.6, 95% CI 2-sided [-13.28 to -3.87]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.3, 95% CI 2-sided [-17.26 to -7.42]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.6, 95% CI 2-sided [-16.51 to -6.78]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -14.3, 95% CI 2-sided [-19.38 to -9.25]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.6, 95% CI 2-sided [-17.53 to -7.70]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1479, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-1.17 to 7.72]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.8382, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-5.16 to 4.19]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.9317, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-4.42 to 4.82]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3169, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-7.29 to 2.37]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.7488, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-5.44 to 3.91]

16. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 54 | 44 | 46 | 39 | 44 | 49 | 40
mmHg | -4.8 (1.09) | -7.4 (1.21) | -6.8 (1.18) | -8.5 (1.29) | -7.8 (1.21) | -6.1 (1.15) | 1.9 (1.27)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-9.98 to -3.40]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.3, 95% CI 2-sided [-12.76 to -5.86]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.6, 95% CI 2-sided [-12.05 to -5.22]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.4, 95% CI 2-sided [-13.92 to -6.79]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.7, 95% CI 2-sided [-13.11 to -6.20]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.4188, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-1.83 to 4.40]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.4255, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-4.62 to 1.95]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.6869, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-3.91 to 2.58]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1678, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-5.77 to 1.01]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3132, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-4.96 to 1.60]

17. Secondary Outcome: Change From Baseline in the 24-36-Hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 24-36-hour mean systolic blood pressure measured at week 8 relative to the 12-hour mean measured at baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-36-hour mean is the average of all measurements recorded from 24 to 36 hours after dosing; the 12-hour mean is the average of the first 12 hours after dosing.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 44 | 45 | 40 | 45 | 49 | 41
mmHg | -9.4 (1.51) | -12.0 (1.64) | -11.5 (1.62) | -14.6 (1.72) | -13.5 (1.62) | -8.9 (1.56) | -1.4 (1.70)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0005, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.0, 95% CI 2-sided [-12.48 to -3.52]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.6, 95% CI 2-sided [-15.24 to -5.93]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.1, 95% CI 2-sided [-14.70 to -5.44]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.2, 95% CI 2-sided [-17.95 to -8.42]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.1, 95% CI 2-sided [-16.74 to -7.48]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.8103, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-4.79 to 3.75]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1702, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-7.57 to 1.34]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2504, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-7.02 to 1.84]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0144, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-10.28 to -1.14]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0402, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-9.06 to -0.21]

18. Secondary Outcome: Change From Baseline in the 24-36-Hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 24-36-hour mean diastolic blood pressure measured at week 8 relative to the 12-hour mean measured at baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-36-hour mean is the average of all measurements recorded from 24 to 36 hours after dosing; the 12-hour mean is the average of the first 12 hours after dosing.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 52 | 44 | 45 | 40 | 45 | 49 | 41
mmHg | -5.6 (1.07) | -7.9 (1.17) | -8.6 (1.15) | -9.5 (1.22) | -7.9 (1.15) | -6.5 (1.11) | -0.4 (1.21)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0014, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.2, 95% CI 2-sided [-8.41 to -2.04]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-10.82 to -4.22]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.2, 95% CI 2-sided [-11.51 to -4.93]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.1, 95% CI 2-sided [-12.49 to -5.72]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.6, 95% CI 2-sided [-10.87 to -4.30]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.5519, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-2.11 to 3.95]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3938, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-4.54 to 1.79]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1949, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-5.21 to 1.07]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0732, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-6.21 to 0.28]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3669, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-4.59 to 1.70]

19. Secondary Outcome: Change From Baseline in the 34-36-Hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 34-36-hour mean systolic blood pressure measured at week 8 relative to the 10-12-hour mean measured at baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-36-hour mean is the average of all measurements recorded from 34 to 36 hours after dosing; the 10-12-hour mean is the average from these 2 hours after dosing.
Time Frame: Baseline and Week 8
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 49 | 43 | 41 | 33 | 42 | 42 | 40
mmHg | -10.1 (1.96) | -11.2 (2.10) | -9.8 (2.15) | -13.5 (2.39) | -11.8 (2.12) | -7.4 (2.12) | -0.9 (2.17)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0019, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.2, 95% CI 2-sided [-14.94 to -3.41]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0008, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.2, 95% CI 2-sided [-16.15 to -4.26]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0040, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.9, 95% CI 2-sided [-14.88 to -2.85]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.6, 95% CI 2-sided [-18.96 to -6.22]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.0004, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.9, 95% CI 2-sided [-16.85 to -4.89]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3499, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-8.39 to 2.98]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2115, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-9.61 to 2.14]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.4279, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-8.34 to 3.54]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.0566, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-12.41 to 0.17]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1435, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-10.30 to 1.50]

20. Secondary Outcome: Change From Baseline in the 34-36-Hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 34-36-hour mean diastolic blood pressure measured at week 8 relative to the 10-12-hour mean measured at baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-36-hour mean is the average of all measurements recorded from 34 to 36 hours after dosing; the 10-12-hour mean is the average from these 2 hours after dosing.
Time Frame: Baseline and Week 8.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Number analyzed (Participants) | 45 | 38 | 39 | 31 | 34 | 33 | 36
mmHg | -0.4 (1.16) | 0.3 (1.26) | 0.9 (1.24) | 0.4 (1.40) | -0.6 (1.34) | 1.9 (1.35) | 2.4 (1.31)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 5 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.1162, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-6.16 to 0.68]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 10 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.2494, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-5.69 to 1.48]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.4247, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.01 to 2.12]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.3007, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-5.79 to 1.80]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.1195, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-6.67 to 0.77]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 5 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.2032, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-5.76 to 1.23]
Statistical Analysis 7: Comparison: Azilsartan Medoxomil 10 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.3787, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-5.27 to 2.01]
Statistical Analysis 8: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.5967, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-4.59 to 2.64]
Statistical Analysis 9: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.4345, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-5.36 to 2.31]
Statistical Analysis 10: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 20 mg QD; Test type: Superiority or Other; p = 0.1954, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-6.24 to 1.28]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 5 mg QD | Azilsartan Medoxomil 10 mg QD | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 20 mg QD | Placebo QD
Serious Adverse Events (participants affected / at risk) | 1/65 | 1/64 | 0/64 | 1/62 | 0/64 | 1/63 | 1/63
Other Adverse Events (participants affected / at risk) | 7/65 | 7/64 | 13/64 | 8/62 | 7/64 | 7/63 | 7/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 5 mg QD (N=65) | Azilsartan Medoxomil 10 mg QD (N=64) | Azilsartan Medoxomil 20 mg QD (N=64) | Azilsartan Medoxomil 40 mg QD (N=62) | Azilsartan Medoxomil 80 mg QD (N=64) | Olmesartan 20 mg QD (N=63) | Placebo QD (N=63)
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive Heart Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal Spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 5 mg QD (N=65) | Azilsartan Medoxomil 10 mg QD (N=64) | Azilsartan Medoxomil 20 mg QD (N=64) | Azilsartan Medoxomil 40 mg QD (N=62) | Azilsartan Medoxomil 80 mg QD (N=64) | Olmesartan 20 mg QD (N=63) | Placebo QD (N=63)
Headache (Nervous system disorders) | 2 | 1 | 7 | 3 | 3 | 5 | 3
Nasopharyngitis (Infections and infestations) | 0 | 3 | 3 | 1 | 3 | 1 | 4
Dizziness (Nervous system disorders) | 1 | 3 | 4 | 2 | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.